CLINICAL TRIAL: NCT05025644
Title: Quantitative Assessment of Hypertrophic Obstructive Cardiomyopathy With Intraoperative Three-dimensional Transesophageal Echocardiography Under Provocative Dobutamine Stress Test
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-5412
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Transesophageal Echocardiography; Dobutamine Stress test
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Lead

STUDY DESIGN:
Intervention Model Description: This is a monocentric Phase IV prospective study that will be conducted on patients undergoing surgical myectomy treatment for HOCM, at Toronto General Hospital, to assess if LVOT gradients may be reproduced with dobutamine provocation test in HOCM patients under general anesthesia.
  The participants in the study will require a standard 2D echocardiography within 6 months pre and post-surgery. Intraoperatively, the patients will be divided into two groups, one with preoperative PG under anesthesia <50mmHg (Group A), and one with preoperative PG under anesthesia ≥ 50mmHg (Group B).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Transesophageal Echocardiogram (TEE) PG under anesthesia <50mmHg (Group A) (Experimental): * Pre-cardiopulmonary bypass (CPB) (pre-myectomy) echocardiographic parameters: PG under DBT stress test at 5, 10, 15 and 20 mcg/kg/min or until a PG ≥ 50mmHg is achieved, will be recorded.
  * Post-CPB (post-myectomy) echocardiographic parameters: PG at DBT peak dose (DBT-pd) will be recorded.
  If LVOT PG post myectomy are >16 mmHg, the surgeon will be advised, for surgical management considerations.
  Interventions: Drug: Pre and post-CPB Drug: Dobutamine Hydrochloride
- Preoperative PG under anesthesia ≥ 50mmHg (Group B) (Experimental): * Pre-cardiopulmonary bypass (CPB) (pre-myectomy) echocardiographic parameters: PG without DBT stress test will be recorded.
  * Post-CPB (post-myectomy) echocardiographic parameters: PG at 5, 10, 15, 20 mcg/kg/min DBT stress test or until the postoperative provocable PG is >16 mmHg will be recorded.
  Interventions: Drug: Post-CPB Drug: Dobutamine Hydrochloride

INTERVENTIONS:
Drug: Pre and post-CPB Drug: Dobutamine Hydrochloride — * Pre-CPB provocation test with DBT stress test will be started (starting at 5 mcg/kg/min, increasing every 3 min, to 10, 15 and 20 mcg/kg/min) until a PG ≥ 50mmHg is achieved (DBT peak dose). The DBT peak dose (DBT-pd) will be recorded.
  * Post-CPB provocation test at the DBT-pd achieved preoperatively.
  Other Names: Transthoracic or 2D Echocardiogram; Transesophageal Echocardiogram (TEE)
  Arms: Preoperative Transesophageal Echocardiogram (TEE) PG under anesthesia <50mmHg (Group A)
Drug: Post-CPB Drug: Dobutamine Hydrochloride — * Pre-CPB no intervention will be required.
  * Post-CPB provocation test with DBT stress test will be started (starting at 5 mcg/kg/min, increasing every 3 min, to 10, 15 and 20 mcg/kg/min) or until postoperative provocable PG is >16 mmHg.
  Other Names: Transthoracic or 2D Echocardiogram; Transesophageal Echocardiogram (TEE)
  Arms: Preoperative PG under anesthesia ≥ 50mmHg (Group B)

SUMMARY:
The objectives of this study are to determine if the left ventricle outflow tract (LVOT) gradients may be reproduced with dobutamine (DBT) provocation test in obstructive HCM patients under general anesthesia and to analyze the change in anatomic LVOT area and pressure gradients (PG) before and after septal myectomy.

If the DBT stress test can reproduce preoperative gradients in HCM patients during septal myectomy surgery, surgeons will have the opportunity to assess the quality of the surgical procedure depending on the obtained gradients with DBT stress test after surgery when gradients can't be reproduced during general anesthesia after myectomy, and decide if further myectomy is required, saving a re-operation on the patient in the future.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is the most common genetic cardiomyopathy. Echocardiography is the noninvasive method of choice for the evaluation of morphologic and functional abnormalities in HCM. It is of paramount importance to distinguish between obstructive or non-obstructive HCM, based on the presence or absence of left ventricle outflow tract (LVOT) gradient using continuous wave Doppler (CWD), under resting and/or provocable conditions. HCM can then be divided into three different subgroups. When the gradient at rest is ≥ 30 mmHg the HCM is considered obstructive (HOCM); when the gradient is <30 mmHg at rest but ≥ 30 mmHg with provocation, the HCM is considered latent obstructive, and finally, non-obstructive occurs when the gradient is < 30mmHg at rest or with provocation.

The gold standard technique to treat symptomatic HOCM is the surgical transaortic septal myectomy, when the resting gradient or the provocable gradient is ≥50 mmHg. Hemodynamic conditions may change and lead to worsening or improvement in LVOT obstruction during general anesthesia. LVOT gradients during surgery should be measured under reproducible conditions possibly mimicking preoperative hemodynamics.

Dobutamine is a well-known inotropic agent, capable to induce sub-aortic gradients in HOCM. The development of a dynamic LVOT gradient during this test is a pharmacological phenomenon with no clinical significance, not been associated with increased frequency of chest pain, shortness of breath or ischemic wall motion abnormalities, because obstruction resolves after termination of dobutamine (DBT) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. HOCM refractory to medical treatment with symptoms like syncope, angina or NYHA functional classes III and IV, with a resting gradient or provocable gradient equal or greater than 50 mmHg, requiring surgical intervention.
2. Absence of other cardiac or systemic diseases capable of producing hypertrophy.
3. Sinus rhythm.

Exclusion Criteria:

1. Patient refusal.
2. Patient unable to give consent.
3. TEE contraindication.
4. Different rhythm than sinus.
5. Other systemic diseases capable of producing hypertrophy.
6. Severe Aortic or coronary artery pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Analyze if TEE immediate post-myectomy LVOT gradients, may be reproduced with provocation dobutamine test in HOCM patients, when compared to TTE LVOT gradients performed within 6 months post-myectomy, to prove septal myectomy efficacy. | Pre-operative up to 6 months, Immediate Intra-operative Pre-myectomy, Immediate Intra-operative Post-myectomy and Post-operative up to 6 months
  The preoperative gradients obtained by TTE, with and without stress test, within 6 months pre-myectomy, will be compared with the intraoperative TEE pre-myectomy gradients at baseline (before and after DBT stress test).
  The post-myectomy TEE gradients (before and after DBT stress test), will be compared with the follow up TTE gradients with and without stress test, performed within 6 months post-myectomy, to assess short term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, Principal Investigator — Sunnybrook Health Science Centre; Azad Mashari, MD, Principal Investigator — University Health Network, Toronto